CLINICAL TRIAL: NCT07333482
Title: Flourish Study: A Randomized, Three-Arm Longitudinal Clinical Study of Microbiome-Guided Interventions in Cesarean-Born Infants
Brief Title: Flourish: Exploring the Early Infant Gut Microbiome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seeding, Inc DBA Tiny Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLOURISH_14952
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Microbiota; Gut Microbiome; Eczema; Microbiome
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full Intervention (Experimental): Participants in the full intervention arm will receive interactive microbiome reports, coaching, personalized recommendations, and educational materials throughout the length of the study.
  Interventions: Dietary Supplement: Tailored Recommendations; Behavioral: Consult Call; Behavioral: Educational Email Series
- Limited Intervention Arm (Experimental): Participants in the limited intervention arm will receive simplified pdf reports with basic probiotic recommendations throughout the study. This arm has the option to participate in report interpretation calls with a Nurse Practitioner.
  Interventions: Dietary Supplement: Tailored Recommendations; Behavioral: Consult Call
- Control Arm (No Intervention): Participants in the control arm will provide the same level of microbiome and survey data as the intervention arms but will not see their results until after the completion of the study.

INTERVENTIONS:
Dietary Supplement: Tailored Recommendations — Recommendations are tailored to the infant's microbiome composition, functional gene profiles (e.g., HMO digestion and SCFA production pathways), age, feeding method, and reported symptoms.
  Guidance may include evidence-based suggestions related to probiotic use, prebiotic intake, and age-appropriate nutritional strategies intended to support healthy gut microbiome development. All recommendations are educational in nature, optional, and provided for consideration by parents or caregivers. No supplements are provided directly as part of the study, and no supplementation is required for study participation.
  Recommendations are updated over time as new microbiome data are collected and are delivered according to study arm assignment. The full intervention arm receives comprehensive, personalized recommendations with interpretive support, while the limited intervention arm receives probiotic recommendations only designed to model a scalable laboratory-developed test (LDT)-style approach.
  Arms: Full Intervention; Limited Intervention Arm
Behavioral: Consult Call — Participants assigned to the full intervention arm will receive scheduled consult calls with a trained microbiome specialist as part of the study intervention. These are conducted remotely and are designed to support participant understanding of microbiome reports, review educational content, and discuss microbiome-informed recommendations in the context of the infant's age, feeding practices, and reported symptoms.
  For participants in the full intervention arm, consult calls may include discussion of microbiome-guided recommendations related to diet, supplementation, and lifestyle factors. Participants in the limited intervention arm may elect to receive a call with a licensed Nurse Practitioner for the purpose of interpreting their static microbiome report only; these calls do not include personalized recommendations or discussion of broader health symptoms. Participants in the control arm do not receive consult calls during the active study period.
  Arms: Full Intervention; Limited Intervention Arm
Behavioral: Educational Email Series — Participants assigned to the full intervention arm will receive a structured educational email series delivered longitudinally over the course of the study. The email series provides evidence-based education on early infant gut microbiome development and its relationship to immune and allergic health outcomes, with links to blog articles summarizing current peer-reviewed research.
  Topics include Cesarean delivery and microbiome seeding, breastfeeding and human milk oligosaccharides, formula selection, probiotic use, antibiotic exposure, gut maturation, introduction of solid foods and allergens, eczema and the atopic march, food sensitivities, environmental microbial exposure, and general strategies to support infant gut health during early life.
  The educational email series is informational only and does not include individualized medical advice. Participants in the limited intervention and control arms do not receive the educational email series during the active study period.
  Arms: Full Intervention

SUMMARY:
The goal of this clinical trial is to learn whether microbiome analysis, education, and personalized recommendations can improve gut health and reduce early markers of immune-related conditions in infants aged 0-3 months delivered via Cesarean section. The study aims to determine whether these interventions can increase beneficial bacteria, decrease C-section-associated microbiome signatures, reduce opportunistic pathogens, and improve functional potential for HMO digestion and SCFA production. The study also seeks to assess whether improvements in microbiome composition are associated with a reduced prevalence of early atopic symptoms.

Researchers will compare three groups: a full intervention arm that receives microbiome reports, coaching, personalized recommendations, and educational materials; a limited intervention arm that receives simplified reports and basic recommendations; and a control arm that receives no results until study completion. This design allows evaluation of both a comprehensive intervention and a more scalable, minimal-results model.

Participants will:

1. Provide six microbiome stool samples over a 24-month period.
2. Provide additional small stool samples at two timepoints for exploratory metabolomic analysis.
3. Receive microbiome reports and guidance according to their assigned study arm.
4. Complete surveys on infant health history, symptoms, diet, and environmental exposures.
5. Participate in standardized eczema assessment(s) administered by a Nurse Practitioner and evaluated by a Pediatric Allergy Specialist if any symptoms are reported.

This study seeks to demonstrate that targeted microbiome support can positively shift gut microbial development in C-section infants and may reduce risks linked to the early stages of the atopic march. Findings may inform scalable strategies for delivering microbiome-based support in early life and improve long-term health outcomes for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Infants are qualified for this study if they are 0 to 3 months of age at time of enrollment.
* Infants must have been delivered via Cesarean delivery (C-section), either scheduled or emergent.
* Infants must have been at least 36 weeks gestation at time of delivery.
* Infants and their caregivers must reside in the United States with a US mailing address.

Exclusion Criteria:

* Infants can not have been given probiotic supplements in their life at recruitment. This includes probiotic powder or supplements or formula with probiotic addition or multivitamin with probiotic addition.
* Twin and multiple birth infants are not accepted in this study.
* Infants cannot have the following existing health conditions:
* Gastrointestinal conditions: Hirschsprung disease, eosinophilic gastrointestinal disorders (EGID) including eosinophilic esophagitis (EoE), necrotizing enterocolitis (NEC), short bowel syndrome (SBS)
* Immune or auto-immune conditions: Severe Combined Immunodeficiency (SCID), human immunodeficiency virus (HIV)), excluding eczema and rashes
* Congenital conditions: cleft lip or cleft palate, congenital heart disease, cerebral palsy, fragile X syndrome, down syndrome, spina bifida, cystic fibrosis, phenylketonuria (PKU), congenital hypothyroidism (CHT), galactosaemia)
* Blood disorders (sickle cell disease, thalassemia, hemophilia)
* Infant or any immediate family member has previously received results from an at-home microbiome stool test (excluding standard clinical diagnostic testing such as stool culture or pathogen testing)

Ages: 0 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Microbiota Composition | 24 months
  Changes in gut microbiota composition, including relative abundance of beneficial bacterial taxa such as Bifidobacterium, assessed using shotgun metagenomic sequencing.
C-Section-Associated Microbiome Signatures | 24 months
  Changes in the relative abundance of microbial taxa and signatures previously associated with Cesarean delivery, assessed longitudinally using shotgun metagenomic sequencing.
Opportunistic and Potentially Pathogenic Microbial Abundance | 24 months
  Changes in the relative abundance of opportunistic and potentially pathogenic microbial taxa over time, assessed using shotgun metagenomic sequencing.
Functional Microbiome Capacity | 24 months
  Changes in microbial functional gene pathways related to human milk oligosaccharide (HMO) digestion and short-chain fatty acid (SCFA) production, assessed using metagenomic functional profiling.
Eczema Incidence / Atopic Symptoms | 24 months
  Incidence of eczema and other early atopic symptoms assessed via parent-reported surveys and standardized eczema assessment when symptoms are reported.

SECONDARY OUTCOMES:
HMO Digestion Functional Capacity | 24 months
  Changes in the abundance of microbial functional gene pathways involved in human milk oligosaccharide (HMO) digestion, assessed using shotgun metagenomic sequencing and functional gene annotation.
  Unit of Measure:
  Relative abundance of HMO digestion-related functional gene pathways
SCFA Production Functional Capacity | 24 months
  Changes in the abundance of microbial functional gene pathways involved in short-chain fatty acid (SCFA) production, assessed using shotgun metagenomic sequencing and functional gene annotation.
  Unit of Measure:
  Relative abundance of SCFA production-related functional gene pathways
Parent-Reported Infant Health Outcomes | 24 months
  Parent-reported infant health outcomes collected via longitudinal surveys, including gastrointestinal symptoms, infections, medication use, and feeding practices.

OTHER OUTCOMES:
Stool Metabolomic Profiles | 24 months
  Description:
  Exploratory characterization of stool metabolite profiles collected at select time points, assessed using untargeted metabolomic analysis.
  Unit of Measure:
  Relative abundance of detected stool metabolites
  Measurement Tool:
  Untargeted stool metabolomics
  Time Frame:
  Select time points through 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Qian Yuan, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Seeding Labs INC, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shao Y, Forster SC, Tsaliki E, Vervier K, Strang A, Simpson N, Kumar N, Stares MD, Rodger A, Brocklehurst P, Field N, Lawley TD. Stunted microbiota and opportunistic pathogen colonization in caesarean-section birth. Nature. 2019 Oct;574(7776):117-121. doi: 10.1038/s41586-019-1560-1. Epub 2019 Sep 18. PMID 31534227
- [Result] Galazzo G, van Best N, Bervoets L, Dapaah IO, Savelkoul PH, Hornef MW; GI-MDH consortium; Lau S, Hamelmann E, Penders J. Development of the Microbiota and Associations With Birth Mode, Diet, and Atopic Disorders in a Longitudinal Analysis of Stool Samples, Collected From Infancy Through Early Childhood. Gastroenterology. 2020 May;158(6):1584-1596. doi: 10.1053/j.gastro.2020.01.024. Epub 2020 Jan 18. PMID 31958431
- [Result] Nieto PA, Nakama C, Trachsel J, Goad D, Soderborg TK, Tan DS, Orlandi A, Yuan Q, Song E, Mueller NT, Mars RA, Hoy CS, Sukhum KV. Improving immune-related health outcomes post-cesarean birth with a gut microbiome-based program: A randomized controlled trial. Pediatr Allergy Immunol. 2025 Sep;36(9):e70182. doi: 10.1111/pai.70182. PMID 40898384